CLINICAL TRIAL: NCT05163600
Title: The Acute Cardiorespiratory Response to Blood-flow Restricted Versus Traditional Exercise Training Regimens (CaRe BFR):4 Randomized Crossover Studies
Brief Title: The Acute Cardiorespiratory Response to Blood-flow Restricted Versus Traditional Exercise Training Regimens (CaRe BFR)
Acronym: CaRe-BFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Christian Clarenbach, PD Dr. med Head of Pneumology, University of Zurich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02038
Record Dates: First submitted 2021-12-03; First posted 2021-12-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: monocenter
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD (Experimental): Diagnosed COPD according to GOLD-guidelines
  Interventions: Other: Blod flow restriction training
- Healthy (Experimental): Age ≥ 18 years Clinically healthy
  Interventions: Other: Blod flow restriction training

INTERVENTIONS:
Other: Blod flow restriction training — includes one strength and one endurance training

SUMMARY:
The investigators hypothesize that BFR exercise regimens result in a different acute cardiorespiratory response pattern compared to traditional exercise regimens. Furthermore, the investigators hypothesize that these patterns differ between healthy participants and participants with COPD.

Regarding secondary objective, the investigators hypothesize that BFR results in lower blood pressure responses compared to traditional exercise training in both healthy and COPD participants.

DETAILED DESCRIPTION:
The investigatorscarry out a monocentric project with 4 randomized crossover studies.

CaRe-BFR Healthy and COPD:

Strength training is performed bilaterally on a Leg Press machine (Leg Press VR2, Cybex International Inc. Medway, MA, USA) using the three set methodology, which is proven to be most effective in enhancing muscle strength.16 Each set is performed to muscular failure, which should be reached within 8-12 repetitions. Training rhythm is set at 1-0-1-0 (i.e. one second for the concentric phase, no pause, one second for the eccentric phase, no pause) and externally paced by a metronome. The training load is 80% of the 1RM. Rest in between sets is 1 minute and participants remain

Strength training BFR is performed bilaterally on a Leg Press machine (Leg Press VR2, Cybex International Inc. Medway, MA, USA) in accordance with evidence-based application guidelines to apply the most effective methodology to enhance muscle strength.17 The exercise consists of a total of 75 repetitions during 4 sets. Training rhythm is set at 1-0-1-0 (i.e. one second for the concentric phase, no pause, one second for the eccentric phase, no pause) and externally paced by a metronome. Set 1 covers 30 repetitions, and the subsequent sets 15 repetitions each. The training load is 30% of the 1RM. Cuffs are mounted bilaterally at the most proximal part of the thigh and inflated to 70% of the individual AOP. Rest in between sets is 1 minute and participants remain seated with the cuffs inflated.

-Endurance is performed bilaterally on a stationary bicycle ergometer (kardiomed 521, proxomed Medizintechnik GmbH, Alzenau, Germany) in an interval setting with loading phases of 1 set with 3 intervals lasting for 2 minutes each; training load is 65% of the peak work rate (PWR). In between the intervals, breaks are standardised to 1 minute. Before the exercise bout, warm-up cycling at 30% PWR for 5 minutes is done to reach a steady state in HR and RER.

Endurance BFR is performed bilaterally on a stationary bicycle ergometer (kardiomed 521, proxomed Medizintechnik GmbH, Alzenau, Germany) in an interval setting with loading phases of 1 set with 3 intervals lasting for 2 minutes and 18 seconds each (matching the overall work performed in EN); training load is 50% of the PWR while limb blood flow is restricted to 50% of the AOP. In between the intervals, breaks are standardised to 1 minute (cuff inflated). Before the exercise bout, warm-up cycling (without BFR) at 30% PWR for 5 minutes is done to reach a steady state in HR and RER.

Measurements:

During exercise, the investigators collect breath-by-breath data (Ergostik, Geratherm Respiratory GmbH, Bad Kissingen, Germany). In addition, continuous SpO2 and HR data via an earlobe probe, and BP response immediately after exercise sets are collected

ELIGIBILITY:
Inclusion and exclusion for the healthy participants are defined by the following criteria.

Inclusion criteria:

* Age ≥ 18 years
* Clinically healthy

Exclusion criteria:

* Physical or intellectual impairment precluding informed consent or protocol adherence
* Non-German speaking (precluding informed consent)
* Pain during exercise of any origin
* Pregnancy
* History of thromboembolic event in the lower extremity
* Resting systolic blood pressure <100 mmHg

Inclusion and exclusion for the COPD participants are defined by the following criteria.

Inclusion criteria:

* Age ≥ 18 years
* Diagnosed COPD according to GOLD-guidelines12

Exclusion criteria:

* Physical or intellectual impairment precluding informed consent or protocol adherence
* Non-German speaking (precluding informed consent)
* Acute or recent (within the last 6 weeks) exacerbation of COPD
* Pain during exercise of any origin
* Pregnancy
* History of thromboembolic event in the lower extremity
* Resting systolic blood pressure <100 mmHg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Within-subject difference in maximal minute ventilation (VE) between BFR and traditional exercise regimens | basline (CPET) 20 min, V1 Training (endurance or strengthwith) with or without BFR 20 min; V2 Training (endurance or strengthwith) with or without BFR 20 min
  investigators will examine VE during strength training and endurance training with and without BFR. Each training sessions will last approximately 20 minutes including baseline CPET.
  There will be no measurements between the trainings. There will be a minimum wait of 48 hours (wash out timne) until training 2 is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Clarenbach, Dr. med, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuhn M, Clarenbach CF, Klay A, Kohler M, Mayer LC, Luchinger M, Andrist B, Radtke T, Haile SR, Sievi NA, Kohlbrenner D. Exploring immediate cardiorespiratory responses: low-intensity blood flow restricted cycling vs. moderate-intensity traditional exercise in a randomized crossover trial. BMC Sports Sci Med Rehabil. 2024 Aug 15;16(1):172. doi: 10.1186/s13102-024-00951-0. PMID 39148127